CLINICAL TRIAL: NCT02181595
Title: Deep Reading as a Contemplative Practice for Women With Primary Ovarian Insufficiency: An Exporatory Pilot Study.
Brief Title: Deep Reading as a Contemplative Practice for Women With Primary Ovarian Insufficiency
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 140139; 14-CH-0139
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2018-03-20

CONDITIONS: Ovarian Insufficiency
Keywords: Reading; FACIT-SP; Primary Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

INTERVENTIONS:
Other: Group reading and discussion

SUMMARY:
Background:

- Women with Primary Ovarian Insufficiency (POI) have ovaries that stopped working normally before they turned 40. This usually causes infertility, which challenges many women with the condition to ask themselves, Why me? This kind of question is about our human existence, or what some call an existential view of life. Researchers have learned that spirituality and finding existential purpose help women with POI. So does meeting other women with the same problem. Researchers want to find new ways to help women with POI cope with it.

Objective:

- To develop and test a practice for women with POI called Deep Reading.

Eligibility:

- Women enrolled in another POI protocol, who can read and speak English.

Design:

* Participants will first have an individual visit or phone call. They will describe spiritual or existential practices they have done. They will also answer questions about spiritual and existential health and daily functioning.
* They will join a group for 6 weekly sessions. Each session will be 60 90 minutes.
* In each group session, a coordinator will teach participants about Deep Reading. They will read a piece of up to 1000 words. They will think about the piece and then talk about it with the group.
* Between sessions, participants will practice Deep Reading at least once for 15 20 minutes on their own. They will check in once with another group member. They will keep a log of these activities.
* After session 3, participants will answer questions online about wellbeing and satisfaction.
* At session 6, participants will answer questions online about wellbeing. They will answer questions about their overall experience.
* One and 3 months after the sessions end, participants will again complete online wellbeing questionnaires and report on their continued practice of Deep Reading.

DETAILED DESCRIPTION:
It is well documented in the literature that women with Primary Ovarian Insufficiency find spirituality a valuable resource for coping with the existential dimension of the diagnosis. This is an exploratory pilot study which examines reading as a contemplative practice to assist these women as they attempt to come to terms with the life altering aspects of living with the diagnosis. In this intervention, that we call Deep Reading, up to 15 participants will engage in six weekly sessions approximately sixty to ninety minutes in length in which they will receive instruction on aspects of Deep Reading, practice Deep Reading and process the experience. Between group sessions participants will be asked to practice Deep Reading on their own and be paired for mutual support and encouragement. For convenience participants will be recruited from among those already enrolled in NICHD Protocol, Ovarian Follicle Function in Patients with Primary Ovarian Insufficiency (91-CH-0127). We will use the FACIT-Sp and satisfaction questionnaires to measure participant response and feasibility for future study.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for this research study, subjects must:

* have previously enrolled in NICHD study 91-CH-0127, Ovarian Follicle Function in Patients with Primary Ovarian Insufficiency
* agree to practice Deep Reading at least once each week outside of group sessions
* agree to respect the privacy and confidentiality of other participants

EXCLUSION CRITERIA:

The following will be excluding from participating in the study:

* those unable to give consent
* those unwilling to participate in 6, 90 minute group sessions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07-02; Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Feasibility based on Acceptability | Recruitment Phase
Feasibility based on Practicality of study | throughout study
Feasibility based on participant opinion | end of study

SECONDARY OUTCOMES:
Changes in FACIT-Sp measure of spiritual well-being | weekly, 1 mon, 3 mon

CONTACTS AND LOCATIONS:
Overall Officials: Margaret F Keil, C.R.N.P., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Puchalski C, Ferrell B, Virani R, Otis-Green S, Baird P, Bull J, Chochinov H, Handzo G, Nelson-Becker H, Prince-Paul M, Pugliese K, Sulmasy D. Improving the quality of spiritual care as a dimension of palliative care: the report of the Consensus Conference. J Palliat Med. 2009 Oct;12(10):885-904. doi: 10.1089/jpm.2009.0142. PMID 19807235
- [Background] Boston P, Bruce A, Schreiber R. Existential suffering in the palliative care setting: an integrated literature review. J Pain Symptom Manage. 2011 Mar;41(3):604-18. doi: 10.1016/j.jpainsymman.2010.05.010. Epub 2010 Dec 8. PMID 21145202
- [Background] Murillo M, Holland JC. Clinical practice guidelines for the management of psychosocial distress at the end of life. Palliat Support Care. 2004 Mar;2(1):65-77. doi: 10.1017/s1478951504040088. PMID 16594236